CLINICAL TRIAL: NCT06473961
Title: An Open, Single-armed, Phase Ib Study to Evaluate the Safety and Efficacy Using Autologous Tumor Infiltrating Lymphocytes Injection (GC101 TIL) in Patients With Non-Small Cell Lung Cancer
Brief Title: A Phase Ib Study of GC101 in NSCLC
Acronym: MIZAR-005
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC101 TIL-NSCLC-Ib
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Participants with advanced NSCLC using cryopreserved GC101 TIL
  Interventions: Biological: Autologous Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Biological: Autologous Tumor Infiltrating Lymphocytes — A tumor sample is resected from each participant and cultured ex vivo to generate tumor infiltrating lymphocytes. After lymphodepletion, patients are infused GC101 TIL followed low-dose PD-1 antibody.
  Other Names: GC101 TIL injection

SUMMARY:
20 participants are expected to be enrolled for the Phase Ib clinical trial，this trail is expected to be finished in 36 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed the informed consent form (ICF) and able to comply with the visits and related procedures specified in the protocol;
* 2. Aged ≥18 years and ≤70 years, regardless of gender;
* 3. Patients with unresectable advanced, recurrent, or metastatic non-small cell lung cancer who are positive for driver genes and have failed after targeted and platinum-containing dual chemotherapy;
* 4. TILs can be isolated from a surgically resectable tumor region: the tissue volume must be >150mm3, and the lesion has not received local treatment (such as radiotherapy, radiofrequency ablation, oncolytic virus, etc.) or progressed after local treatment;
* 5. There are still at least 1 measurable lesion (according to RECIST1.1 criteria [see Appendix 4]) even after TIL sampling and resection of surgically resectable tissue;
* 6. ECOG performance status 0-1;
* 7. Expected survival time >3 months;
* 8. With sufficient hematology and end-organ function as defined by the following laboratory test results, the test results must be completed and issued within 7 days before tumor tissue collection:

  * White Blood Cell (WBC)≥2.5×10^9/L#
  * Absolute Lymphocyte Count (ANC)≥1.5×10^9/L;
  * Absolute Lymphocyte Count(ALC)≥0.7×10^9/L;
  * Platelet≥100×10^9/L#
  * International Normalized Ratio#INR#≤1.5×ULN;
  * Activated Partial Thromboplastin Time#APTT#≤1.5×ULN;
  * Serum Creatinine (Scr)≤1.5mg/dL (or 132.6μmol/L) or Creatinine
  * Clearance≥60mL/min
  * Urinalysis: urine protein less than 2+, or 24-hour urine protein <1g;
  * Alanine aminotransferase(AST/SGOT) ≤3×ULN;
  * Alanine aminotransferase (ALT/SGPT) ≤3×ULN;
  * Total Bilirubin(TBIL)≤1.5×ULN#
* 9. * Premenopausal women who have not undergone sterilization surgery must agree to use effective contraception measures from the start of study treatment (preconditioning) to one year after cell infusion, and the serum pregnancy test during the screening period must be negative; *Men who have not undergone sterilization surgery must agree to use effective contraception measures from the start of study treatment (preconditioning) until one year after cell infusion;
* 10. No absolute or relative contraindications for surgery;
* 11. Any melanoma treatment methods, including radiotherapy, chemotherapy, endocrine therapy, targeted therapy, immunotherapy, tumor embolization, or traditional Chinese medicine/herbal medicine treatment with anti-tumor indications, must be stopped 28 days before infusion. If a small molecular targeted drug was used in the previous treatment, the withdrawal time can be shortened to 5 half-lives of the drug used;
* 12. Good compliance and able to adhere to the study visit plan and other agreement requirements.

Exclusion Criteria:

* 1. More than 5-line system therapy had been used in previous 3 years before screening period.
* 2. Participation in a clinical trial of another drug or biologic therapy or receipt of a comparable cellular therapy within 28 days prior to infusion;
* 3. Combination of 2 or more malignant tumors, except: Eradicated malignant tumors that have been inactive for ≥5 years prior to study entry and are at minimal risk of recurrence; adequately treated non-melanoma skin cancer or malignant nevus of freckle-like nevus without evidence of disease recurrence; adequately treated carcinoma in situ without evidence of disease recurrence;
* 4. Has received live attenuated vaccination after signing informed consent or is scheduled to receive it during the study;
* 5. Has not recovered from a prior procedure or treatment-related adverse reaction to ≤ grade 1 nci ctcae 5.0 (except for toxicities such as alopecia, etc., which in the judgment of the investigator pose no safety risk);
* 6. Known history of allergy to streptomycin, ciprofloxacin, or micafungin or allergy to any component of the infused product formulation;
* 7. Uncontrolled co-morbidities including, but not limited to, uncontrolled arterial hypertension (systolic blood pressure ≥160 mmhg and/or diastolic blood pressure ≥100 mmhg) even with standardized treatment or any unstable cardiovascular disease including transient ischemic attack, cerebrovascular accident, myocardial infarction, unstable angina pectoris within 6 months prior to enrollment; new york heart association ( nyha class iii or iv congestive heart failure with an ejection fraction <50%; or severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias, degree ii-iii atrioventricular block, etc., requiring clinical intervention; ecg results showing clinically significant abnormalities or a qtcf ≥450ms (if the first test is abnormal, it may be retested at least 5 minutes apart twice and the combined result/mean value to determine eligibility) ;
* 8. Patients with esophageal or gastric varices that require immediate intervention (e.g., taping or sclerotherapy) or are considered to be at high risk for bleeding based on the opinion of the investigator or consultation with a gastroenterologist or hepatologist, have evidence of portal hypertension (including splenomegaly detected on imaging), or have a prior history of variceal bleeding must have undergone endoscopic evaluation within 3 months prior to enrollment;
* 9. Uncontrolled metabolic disorders, such as diabetes mellitus known to be uncontrolled, or other non-malignant organ or systemic diseases or secondary reactions to cancer, and which can lead to higher medical risk and/or uncertainty in survival evaluation;
* 10. Hepatic encephalopathy, hepatorenal syndrome or child-pugh class b or more severe cirrhosis, liver failure;
* 11. Comorbidity with other serious organic or psychiatric disease;
* 12. Have an active systemic infection requiring treatment with positive blood cultures or imaging evidence of infection, including but not limited to active tuberculosis;
* 13. Be hiv-positive, have a positive serologic test for syphilis, or have clinically active hepatitis a, b, or c, including viral carriers: Hepatitis b, excluding those who are HBsAg-positive; hepatitis c, excluding those who are HCVAb-positive;
* 14. Active autoimmune diseases that still require systemic steroid hormones or other immunosuppressive drugs during the screening period (greater than 10 mg/ day of prednisone or equivalent doses of other hormones);
* 15. Any nci ctcae5.0 immune-related adverse effect (irae) grade ≥ 3 during any prior period of immunotherapy receipt;
* 16. History of organ allograft, allogeneic stem cell transplantation and renal replacement therapy; History of allogeneic t-cell and nk-cell therapy;
* 17. Pulmonary fibrosis, interstitial lung disease (both past history and current), and acute lung disease; Patients with obstructive or restrictive lung disease with FEV1(forced expiratory volume in 1 second) of lung function ≤70%;
* 18. Clinically uncontrollable third space effusions, such as pleural and abdominal effusions that cannot be controlled by drainage or other means prior to enrollment;
* 19. Patients with clinically symptomatic central nervous system metastases (e.g., cerebral edema, need for hormonal intervention, or progression of brain metastases). Patients with prior treatment for brain metastases, such as clinical stability (mri) that has been maintained for at least 2 months and who have discontinued systemic hormone therapy (dose >10 mg/day prednisone or other equipotent hormone) for >4 weeks may be included;
* 20. Women who are pregnant or breastfeeding;
* 21. If the investigator believes that other circumstances are not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to Day 28
  Incidence of adverse events associated with GC101 TIL retransfusion
Objective Response Rate | 18 weeks
  Proportion of subjects in total cases in complete or partial response (RECIST v1.1 criteria)

SECONDARY OUTCOMES:
Adverse Events | Maximum 360 days
  Incidence of adverse events associated with GC101 TIL retransfusion
Objective Response Rate | Maximum 36 months
  Proportion of subjects in total cases in complete or partial response (RECIST v1.1 criteria) during the study
Best overall response | Maximum 36 months
  Optimal efficacy recorded from the start of treatment until disease progression or relapse (RECIST v1.1 and iRECIST)
Disease Control Rate | Maximum 36 months
  Evaluate the efficacy endpoints of DCR by the investigator with RECIST v1.1 and iRECIST
Progression-Free Survival | Maximum 36 months
  Evaluate the efficacy endpoints of PFS by the investigator with RECIST v1.1 and iRECIST
Duration of Response | Maximum 36 months
  Evaluate the efficacy endpoints of DOR by the investigator with RECIST v1.1 and iRECIST
overall survival | Maximum 36 months
  Evaluate the efficacy endpoints of OS

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No